CLINICAL TRIAL: NCT04847882
Title: Sleep Disorders in Patients Aged From 6 to 17 With Cystic Fibrosis: a Single-center Case-control Study at Strasbourg University Hospital
Brief Title: Case-control Study of Sleep Disorders in Children With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8228
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cystic Fibrosis; Sleep Disorder
Keywords: Children; Case control study
MeSH Terms: conditions — Cystic Fibrosis; Sleep Wake Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis, children from 6 to 17.: This group is made up of children with cystic fibrosis followed at the Strasbourg pediatrics CRCM, aged from 6 to 17 years old, not hospitalized at the time of inclusion, without any other criterion prejudging the seriousness of the pathology.
  Interventions: Behavioral: Questionnaire
- Control group, children from 6 to 17.: This group is the control group. It is made up of children consulting in pediatric surgical emergencies, aged 6 to 17 years. Surgical emergencies were chosen because it is a point of consultation, rather accidental, where sleep has often not been impacted in the previous months and where the frequency of chronic pathology is not higher than the general population.
  An other criteria is that these children are accompanied by at least one of their parents and that they can read and understand French well.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire submitted to the parents of children with cystic fibrosis aged 6 to 17 years and to controls in order to assess and compare the prevalence of sleep disorders and their main non-respiratory causes

SUMMARY:
Our primary purpose is to compare the prevalence of sleep disorders in children aged 6 to 17 with cystic fibrosis versus controls with a Sleep disorder screening score, the SDSC. Our hypothesis is that patients aged 6 to 17 with cystic fibrosis have a higher prevalence of sleep disturbances than the general population of the same age group.

Our secondary hypothesis is that these sleep disorders are mixed and that there are non-respiratory causes, sometimes modifiable by simple non-medical treatment and that's why our secondary purpose is to identify the responsible factors, in particular non-respiratory factors in the 2 groups and to compare them.

ELIGIBILITY:
Inclusion criteria for the case group :

* Cystic fibrosis followed at the pediatric (Centre de Ressources et de Compétences de la Mucoviscidose) in Strasbourg
* Aged from 6 to 17 years old
* Non hospitalized
* Able to read and understand French language
* Accompanied by at least one of his parents

Inclusion criteria for the control group :

* Emergency surgical consultation
* Aged from 6 to 17 years old
* Non hospitalized
* Able to read and understand French langage
* Accompanied by at least one of his parents

Exclusion criteria:

* Children under 6 years old
* Children over 17 years old
* Children and parents who don't understand or can't read French language
* Hospitalized children
* Children unaccompanied by their parents

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 6 to 17 years with cystic fibrosis for the case group and children with an emergency surgical consultation for the control group
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Questionnaire SDSC | 15 minutes
  The specific measure for our first purpose is a validated questionnaire called SDSC for "Sleep Disturbance Scale for Children"

SECONDARY OUTCOMES:
Questionnaire SDSC | 15 minutes
  Questions about sleep and life hygiene, various pathologies to highlight modifiable non-respiratory factors of sleep disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaire de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided